CLINICAL TRIAL: NCT01544855
Title: Does Incorporation of EPA and DHA in Lipoproteins Differ According to Apolipoprotein E Genotype?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Mélanie Plourde, Assistant Professor, Université de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Centrum
Record Dates: First submitted 2012-02-24; First posted 2012-03-06 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Healthy
Keywords: Health young participants
MeSH Terms: interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- APOE4 carriers (Experimental): The results obtained for APOE4 carriers will be compared to the one obtained from APOE4 non-carriers. Carriers are defined as being at least carrier of one APOE4 allele.
  Interventions: Dietary Supplement: omega-3 fatty acids

INTERVENTIONS:
Dietary Supplement: omega-3 fatty acids — Participants will take 700 mg/d of EPA and 500 mg/d of DHA as ethyl esters for one month (Ocean Nutrition, Dartmouth, NS) which is about 10 times the current estimated intake of young adults (21). This corresponds to one capsule with breakfast and one capsule with diner.

SUMMARY:
Genetics and nutrition both clearly affect the risk of Alzheimer's disease (AD) in the elderly. Apolipoprotein E (APOE4) is the most important known genetic risk for AD and is prevalent in 20-25% of Canadians, but at present, knowing an individual's ApoE genotype does not help the diagnosis, treatment or prevention of AD. Furthermore, fish intake containing docosahexaenoic acid (DHA, 22:6 omega-3) and eicosapentaenoic acid (EPA, 20:5 omega-3) may be incorporated as a prevention strategy for lowering the risk of AD. However, fish intake seems not to protect APOE4 carriers from developing AD. One explanation as to why APOE4 carriers may not benefit from fish intake is potentially linked with imbalances in omega-3 fatty acid metabolism. The investigators recently reported that after 3g/d of EPA+DHA for 6 weeks, increases in the two fatty acids was less for carriers resulting in a significant gene-by-diet interaction. ApoE is a component of lipoproteins and ApoE genotypes modulate the fasting lipoprotein response to fish-oil supplementation. Therefore, the investigators hypothesis is that APOE4 genotype is associated with imbalances in lipoprotein concentrations which has the consequence to be associated with imbalances in EPA and DHA transport. The investigators will recruit and test 100 healthy young adults since at older ages carriers of ApoE4 usually take medication altering their lipoprotein profile. They will receive an EPA + DHA supplement for one month. This period was chosen because the 3 class of lipoproteins (VLDL, LDL and HDL) have different concentrations in TG, phospholipids and cholesteryl esters and to fully investigate lipoprotein fatty acid changes, one month of supplementation is needed to change EPA and DHA in all lipid classes. The investigators will monitor the distribution of EPA and DHA in the lipoproteins over a one month supplementation with fish oil and the investigators will separate the investigators groups by APOE4 carriers and non-carriers.

ELIGIBILITY:
Inclusion Criteria:

* Fifty healthy men and fifty healthy women aged between 20-35 y old will be recruited.

Exclusion Criteria:

* Tobacco
* Medication (except for oral contraceptives)
* EPA+DHA supplements
* Cancer
* Recent major surgery (< 2 years)
* Ongoing or past severe drug or alcohol abuse
* History of psychiatric difficulties or depression
* Allergy to seafood
* Elite level of physical training
* Pregnancy and breastfeeding

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Distribution of EPA and DHA in lipoproteins by APOE genotype | Once each week for 28 days
  We will measure % and concentration of EPA and DHA in VLDL, HDL and LDL to evaluate how these fatty acids are transported in the blood and whether APOE genotype changes the distribution of these fatty acids.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de recherche sur le vieillissement, Sherbrooke, Quebec, Canada

REFERENCES:
- [Derived] Conway V, Allard MJ, Minihane AM, Jackson KG, Lovegrove JA, Plourde M. Postprandial enrichment of triacylglycerol-rich lipoproteins with omega-3 fatty acids: lack of an interaction with apolipoprotein E genotype? Lipids Health Dis. 2014 Sep 16;13:148. doi: 10.1186/1476-511X-13-148. PMID 25227179